CLINICAL TRIAL: NCT01927328
Title: An Pilot Study to Assess the Efficacy of Intravenous Iron Isomaltoside 1000 (Monofer®) in the Management of Anaemia Associated With the Palliative Management of Oesophagogastric Adenocarcinoma
Brief Title: Iron Replacement in Oesophagogastric Neoplasia
Acronym: IRON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12GA029; 2013-000209-22 (EudraCT Number)
Record Dates: First submitted 2013-08-05; First posted 2013-08-22 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Anemia; Esophageal Cancer; Gastric Cancer
Keywords: Adenocarcinoma; Anemia; Palliative therapy; Palliative care; Palliative treatments; Chemotherapy; Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Anemia; Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma | interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard Care as determined by the clinical team
- Iron isomaltoside 1000 (Active Comparator): Intravenous Iron Isomaltoside 1000 (Monofer®)will be administered in line with the summary of product characteristics.
  Interventions: Drug: Iron isomaltoside 1000

INTERVENTIONS:
Drug: Iron isomaltoside 1000
  Other Names: Monofer®
  Arms: Iron isomaltoside 1000

SUMMARY:
40 eligible patients with confirmed esophageal or gastric adenocarcinoma and anemia will be randomized to a control or intervention group for management of this anemia. The control group treatment will consist of standard treatments as governed by the clinical team (eg oral iron, blood transfusions) whilst the intervention group will be treated with intravenous iron III isomaltoside (Monofer ®).

It is hypothesized that intravenous iron supplementation is more efficacious than standard therapies.

DETAILED DESCRIPTION:
Anemia is a common problem to affect patients diagnosed with esophageal or gastric cancer. This anemia is thought to be secondary to blood loss from the tumor, poor oral intake resulting from symptoms of the tumor, and impaired iron absorption secondary to neoplasia induced inflammatory processes.

Patients undergoing palliative chemotherapy for esophageal or gastric adenocarcinoma are thus prone to development or exacerbation of anemia during their chemotherapy, as this tumor is remains in situ.

Anemia results in symptoms such as shortness of breath, fatigue, lethargy and chest pain, which can all affect quality of life. Oral iron and blood transfusions are the current mainstay of treatment for the condition, yet both have their disadvantages. Oral iron is often poorly tolerated due to side effects including constipation, diarrhea, abdominal pain and nausea. Blood transfusions can also be administered but expose the patient to other risks including infection and transfusion associated reactions. In order to overcome these issues, intravenous iron preparations have been developed and have improved in safety.

This is a single-center, randomized, open label, clinical trial, which looks to investigate the efficacy of intravenous iron is in the treatment of anemia in patients with a diagnosis of esophageal or gastric adenocarcinoma.

Patients will be randomized to receive intravenous iron III isomaltoside (treatment group) or standard therapies decided by the clinical team (control). The outcomes reviewed will include the amount and frequency of blood transfusions received, changes in patient blood profiles and most importantly, patient quality of life scores. Patients will be followed from the start of their chemotherapy until the beginning of the third cycle.

The primary hypothesis to be tested is that intravenous iron will increase quality of life by reducing the symptoms of anemia. We also hypothesize that there will be a decrease in blood transfusion rate in this group and improved changes in hemoglobin and hematinics.

This is designed as a pilot study to determine the feasibility of a larger trial. Randomization will be performed using random allocation of opaque envelopes. All data will be confidentially recorded, as will drug reactions and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing/able to give informed consent for study participation.
* Male or Female, aged 18+
* Anemic with hemoglobin values <13 g d/L for males & < 11.5 g/dL for females.
* Diagnosed with histologically proven esophageal,gastric or Gastro-esophageal Junctional adenocarcinoma.
* Treatment selected is palliative chemotherapy.
* Medically fit for initiation of palliative chemotherapy.
* Able (in the Investigators opinion) & willing to comply with all study aspects.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Patients who following investigation do not have a histological diagnosis of upper GI adenocarcinoma
* Female participants who are pregnant, lactating or planning a pregnancy during the course of the study.
* Patients with evidence of iron overload or disturbances in utilization of iron as stated in the product Summary of Product Characteristics.
* Known hematological disease that, in the investigators opinion would confound any changes in blood results.
* Features necessitating urgent surgery.
* Previous allergy to intravenous iron or related iron products.
* Patients who are unable to consent.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Donation of blood during the study.
* Prisoners and minors (<18 years).
* Non-iron deficiency anaemia (e.g. haemolytic anaemia).
* Hypersensitivity to the active substance or to any of the excipients.
* Patients with a history of asthma, allergic eczema or other atopic allergy.
* Decompensated liver cirrhosis and hepatitis.
* Rheumatoid arthritis with symptoms or signs of active inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin differences between groups | 8 months
  This will govern the magnitude of treatment effect, and hence aid design of a larger study.

SECONDARY OUTCOMES:
Differences in quality of life | 0-14 weeks
  To compare quality of life scores as determined by the EQ-5D and FACT-An questionnaires between treatment groups
Number of allogenic red blood cell transfusions administered | 0-14 weeks
  To investigate if the number of units transfused per participant, the number of participants whom received a blood transfusion and the total number of units of blood transfused differs between the two study arms. This period monitored will begin at enrolment into the study, and cease at the start of the third cycle of chemotherapy
Differences in hematinic markers. | 0 - 14 weeks
  To evaluate if hematinic markers (ferritin, iron, transferrin, transferrin) differ between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Barrie D Keeler, FRCS, Principal Investigator — University of Nottingham; Austin G Acheson, MD FRCS, Study Chair — University of Nottingham
Locations (1):
- Nottingham Univeristy Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom